CLINICAL TRIAL: NCT00427739
Title: Pilot Study of Data Collection During Computerized Tomography (CT) to Determine Accurate Flow Rates for Axial Flow Ventricular Assist Device (VAD) Patients
Brief Title: Data Collection During CT for Axial Flow VADs
Status: Completed | Type: Observational
Sponsor: Subha Raman (Other)
Responsible Party: Sponsor-Investigator, Subha Raman, Professor of Medicine, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2005H0200
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: Axial Flow Ventricular Assist Device; Cardiac CT; Stage IV heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCT exam
  Interventions: Procedure: Cardiac CT

INTERVENTIONS:
Procedure: Cardiac CT — 64 slice spiral computerized tomography

SUMMARY:
At present, there is not accurate way to determine specific flow rates for axial flow ventricular assist devices (VADS). If a right heart cath is needed for these patients for clinical purposes, they will also undergo a cardiac CT scan while the pulmonary artery catheter is in place. It is possible to visualize the flow rates of axial flow VAD's and determine a more accurate rate per specific patient.

Data Analyzed with following results:

Article in Press for Cardiopulmonary Support and Physiology, results state "Pairwise comparison of calculated output from left ventricular assist devices is feasible using first pass dynamic computed tomography test bolus technique versus thermodilution output measurements yielded good agreement (P=.03). The output calculated using dynamic CT underestimated the thermodilution output measurement by 0.54+ 0.37 L/min (95% confidence interval 0.66-0.94).

DETAILED DESCRIPTION:
Description as listed in Summary. The hemodynamic data collected along with pump parameters may help determine more accurate flow rates specific to each patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with implanted left ventricular assist devices referred for CT scans
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
data collection to help determine better clinical evaluation | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Sun, MD, Principal Investigator — Ohio State University, Division of Cardiothoracic Surgery
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States